CLINICAL TRIAL: NCT06545760
Title: Admission to the Kangaroo Mother Care Ward and Maternal Postpartum Depression: a Randomized Controlled Trial
Brief Title: Admission to Kangaroo Mother Care (KMC) Ward and Maternal Postpartum Depression
Acronym: KMC PPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); University of Zambia (Other); University of Cincinnati (Other); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Albert Manasyan, MD, MPH, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UAB-300012872; TTS-2404-65126 (Other Grant/Funding Number: Grand Challenges Canada); 000544699 (Other: UAB OSP)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Low Birth Weight; Kangaroo Mother Care; Postpartum Depression; Neurodevelopmental Outcome; Pre-Term
Keywords: Low resource setting; Kangaroo Mother Care; Paternal depression; Cost-effectiveness
MeSH Terms: conditions — Depression, Postpartum; Premature Birth | interventions — Kangaroo-Mother Care Method; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Admission to Kangaroo Mother Care (KMC) ward for > 2 days after discharge from NICU (Experimental): Following discharge from the neonatal intensive care unit (NICU), preterm mothers and their infants will be discharged to an inpatient kangaroo mother care (KMC) ward for greater than 2 days for continued support.
  Interventions: Behavioral: Kangaroo mother care (KMC) support for > 2 days
- Admission to Kangaroo Mother Care (KMC) ward for < 2 days after discharge from NICU (Placebo Comparator): Following discharge from the neonatal intensive care unit (NICU), preterm mothers and their infants will be discharged to an inpatient kangaroo mother care (KMC) ward for less than 2 days for continued support.
  Interventions: Behavioral: Kangaroo mother care (KMC) support for < 2 days

INTERVENTIONS:
Behavioral: Kangaroo mother care (KMC) support for > 2 days — Admission to the kangaroo mother care (KMC) ward with continued support of kangaroo mother care, breastfeeding, and preterm infant care for greater than 2 days prior to discharge home
  Other Names: Extended kangaroo mother care (KMC)
  Arms: Admission to Kangaroo Mother Care (KMC) ward for > 2 days after discharge from NICU
Behavioral: Kangaroo mother care (KMC) support for < 2 days — Admission to the kangaroo mother care (KMC) ward with continued support of kangaroo mother care, breastfeeding, and preterm infant care for less than 2 days prior to discharge home
  Other Names: Routine kangaroo mother care (KMC)
  Arms: Admission to Kangaroo Mother Care (KMC) ward for < 2 days after discharge from NICU

SUMMARY:
The goal of this clinical trial is to learn if extended admission to the Kangaroo Mother Care (KMC) ward helps to prevent postpartum depression in mothers of low birthweight infants in a low-resource setting whose newborns were admitted to the neonatal intensive care unit (NICU) more than standard of care KMC. The main questions it aims to answer are:

* Does longer KMC decrease the incidence of postpartum depression in mothers of low birthweight infants in a low-resource setting?
* Does longer KMC improve neurodevelopmental outcomes of low birthweight infants at 6, 12, and 18 months in a low-resource setting?
* What are the barriers to practicing KMC in low birthweight infants following hospital discharge in a low-resource setting?
* What is the prevalence of paternal depression in a low resource setting?
* Is it cost effective to admit preterm mother-infant dyads to the KMC ward following NICU discharge?

Researchers will compare (extended admission to the KMC ward) to (standard of care KMC) to see if extended KMC decreases PPD in mothers of preterm infants in low-resource settings.

Participants (infants) will:

* At time of discharge from the NICU, when clinically stable, spend either < 2 days in the KMC ward with their mothers or spend longer in the KMC ward until discharge.
* Return to clinic at routine follow-up visits (at 2 weeks and at 6-8 weeks) where mothers will be screened for postpartum depression and fathers will be screened for depression.
* Return to clinic for neurodevelopmental screening at 6, 12, and 18 months where mothers will be screened for postpartum depression and perceived social support and fathers will be screened for depression.

DETAILED DESCRIPTION:
The overarching objective is to determine whether initiation of Kangaroo Mother Care (KMC) at the neonatal intensive care unit (NICU) followed by admission to the KMC ward for continued support for more than 2 days before discharge home reduces maternal postpartum depression (PPD) and other maternal and infant adverse outcomes in low-resource settings. The central hypothesis is that NICU KMC plus admission of mother-infant (preterm) dyads to the KMC ward following NICU discharge for more than 2 days will reduce the risk of maternal PPD as compared to NICU KMC followed by admission of the mother-infant dyad to the KMC ward for up to 2 days only.

The study aims are:

Aim 1: To determine the effect of admission of mother-infant dyads to the KMC ward following NICU for more than 2 days on maternal PPD at 2-weeks, 6-8 weeks, 6 months, and 12 months.

Aim 2: To determine the effect of admission of mother-infant dyads to the KMC ward on infant's developmental outcomes at 6-,12-, and 18 months of age.

Aim 3: To characterize the feasibility and barriers to uptake of KMC at the hospital and following discharge.

Aim 4: To determine the prevalence of paternal depression.

Aim 5: To estimate the cost and effectiveness of admission of low birthweight infants to the KMC ward:

1. Estimate costs from a health systems perspective and explore cost drivers of KMC and NICU care for low birthweight newborns
2. Assess out-of-pocket expenditure incurred by households due to admission of low birthweight infants to the KMC and NICU
3. Estimate the incremental cost-effectiveness of screening for postpartum depression among women with low birthweight infants admitted to the KMC compared to the status quo

Study design This study is a randomized controlled trial of newly delivered women whose preterm newborns have been admitted to the neonatal intensive care unit (NICU) with admission to the Kangaroo Mother Care (KMC) ward for up to 2 days (control) or with admission to the KMC ward for more than 2 days (intervention) prior to discharge home. The study will enroll a total of 1908 study participants from both study arms pulled from 612 mothers (aim #1), 612 infants (aim #2), 72 participants for in-depth interviews (aim #3), and 612 fathers (aim #4).

ELIGIBILITY:
Inclusion Criteria:

-AIM #1-2 and #5

Mothers to newborns who are:

1) Birthweight between 1000-2000gm 2) Admitted to the Women and Neonates Hospital-University Teaching Hospital Neonatal Intensive Care Unit (WNH-UTH NICU) (>48hrs) 3) Stable preterm eligible for continuing kangaroo mother care (KMC) in the NICU or NICU discharge 4) 18+ years of age (Mother) 5) Residing within Lusaka with no intensions to relocate in the coming 12 months

* AIM #3

  1. Parents (mothers and fathers) whose newborn has been enrolled in the study
  2. Trusted family member or friend of the mother whose newborns is enrolled into the study
  3. 18+ years of age
* AIM # 4:

  1. Fathers whose newborn has been enrolled into the study
  2. 18+ years of age (father)

Exclusion Criteria:

* AIM #1-2 and #5

  1. Mothers who are on treatment for depression and/or anxiety
  2. Mothers who did not consent
* AIM #3

  1) Family members of parents who do not consent to study participation
* AIM # 4:

  1. Fathers who are on treatment for depression and/or anxiety
  2. Fathers who did not provide informed consent

Ages: 1 Day to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1908 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Mothers with Postpartum Depression (PPD) | 8 weeks
  Score on Edinburgh Postnatal Depression Scale (EPDS) screening tool obtained by interview with mother. This screening tool is a 10-question tool validated for use among pregnant women in low resource countries. It can be used for screening of perinatal depression, beginning from antenatal period up to 6-8 weeks postnatal age. Each question is scored between 0-3, the highest cumulative score being 30. Cut-off score for mothers with suspected postpartum depression (PPD) will be 11. All mothers who screen 11+ will be categorized to have PPD, all mothers scoring below 11 will be categorized as negative for PPD.

SECONDARY OUTCOMES:
Percentage of Mothers with Postpartum Depression (PPD) | 2 weeks, 6 months, 12 months
  Score on Edinburgh Postnatal Depression Scale (EPDS) screening tool obtained by interview with mother. This screening tool is a 10-question tool validated for use among pregnant women in low resource countries. It can be used for screening of perinatal depression, beginning from antenatal period up to 6-8 weeks postnatal age. Each question is scored between 0-3, the highest cumulative score being 30. Cut-off score for mothers with suspected postpartum depression (PPD) will be 11. All mothers who screen 11+ will be categorized to have PPD, all mothers scoring below 11 will be categorized as negative for PPD.
Hours spent practicing Kangaroo Mother Care (KMC) in the neonatal intensive care unit (NICU) | 2 weeks
  Time in hours and minutes spent practicing kangaroo mother care (KMC) per day by the mother obtained by interview with mother.
Hours spent practicing Kangaroo Mother Care (KMC) in the KMC Ward | 2 weeks
  Time in hours and minutes spent practicing kangaroo mother care (KMC) per day by the mother obtained by interview with mother.
Hours spent practicing Kangaroo Mother Care (KMC) at home | 2 weeks, 8 weeks, 6 months, 12 months
  Time in hours and minutes spent practicing kangaroo mother care (KMC) per day by the mother obtained by interview with mother.
Time of initiation of breastfeeding | 2 weeks
  Time in hours and minutes after delivery, when infant is initially put to breast for feeding
Number of months breastfeeding | 8 weeks, 6 months, 12 months
  Number of months of any breastfeeding reported by the mother in an interview
Number of barriers to kangaroo mother care (KMC) initiation at the birth hospital | 12 months
  A pre-defined set of questions will be asked to all the mothers to determine the barriers contributing to kangaroo mother care (KMC) initiation at the birth hospital. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Number of barriers to kangaroo mother care (KMC) initiation at home | 12 months
  A pre-defined set of questions will be asked to all the mothers to determine the barriers contributing to kangaroo mother care (KMC) initiation at home. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Average Infant/child developmental assessment | 6 months,12 months, 18 months
  Score on "Ages and Stages Questionnaire" (ASQ) obtained by interview with parent developmental assessment tools which scores items (Y = 10, Sometimes = 5, Not Yet = 0) in areas of Communication, Gross motor, Fine Motor, Problem Solving and Personal-Social. Scoring of items are totaled and placed on a graph indicating cut off score. If score is above cut-off, the child's development appears to be on schedule; near the cutoff, may provide learning activities and monitor; and below cutoff, requiring further assessment.
  6-month cutoffs (Communication 29.65; Gross Motor 22.25; Fine Motor 25.14; Problem Solving 27.72 and Personal-Social 25.34); 12-month cutoffs (Communication 15.64; Gross Motor 21.49; Fine Motor 34.50; Problem Solving 27.32 and Personal-Social 21.73); 18-month cutoffs (Communication 13.06; Gross Motor 37.38; Fine Motor 34.32; Problem Solving 25.74 and Personal-Social 27.19).
Average weight in grams | birth, up to 8 weeks, 6 months, 12 months, 18 months
  Weight in grams, weighed on a digital scale
Average length in centimeters (cm) | birth, up to 8 weeks, 6 months, 12 months, 18 months
  Length in centimeters, top of head to heel, measured with paper tape measure
Average head Circumference in centimeters (cm) | birth, up to 8 weeks, 6 months, 12 months, 18 months
  Head Circumference in centimeters (cm), occipital-frontal, measured with paper tape measure
Percentage of all cause 28-day neonatal mortality | 28 days
  Report of neonatal vital status within 28 days, obtained in maternal interview
Percentage of neonatal morbidity | 28 days
  Report of neonatal health status, obtained in maternal interview (e.g., neonatal sepsis, diarrhoea, breathing difficulties)
Percentage of infant readmission to facility | 18 months
  Neonatal rehospitalization after initial discharge from the hospital assessed by maternal interview or medical records documentation
Percentage of infant mortality | 18 months
  Documentation of or report of infant death, assessed through medical records or maternal interview
Percentage of infant morbidity | 18 months
  Report of infant morbidity, assessed through maternal interview (e.g., diarrhoea, pneumonia, sepsis, respiratory infections)
Percentage of vaccine adherence | 12 months
  Report of infant's adherence to the required vaccinations per national guidelines in Zambia through maternal interview -
  Bacille Calmette-Guérin (BCG) - at birth Polio (Oral Polio Virus 0, 1, 2, 3) - birth, 6, 10, and 14 weeks Diphtheria, tetanus, whooping cough (pertussis) or DTP, polio, hepatitis B and Haemophilus influenzae type b (Hib) - DPT-HepB-HiiB (1, 2, 3) - at 6, 10, and 14 weeks Measles - at 9 and 18 months Rotavirus 1, 2 - at 6 and 14 weeks Preumococcal Vaccine (PCV) 1, 2 - at 6, 10, and 14 weeks
Number of barriers to practicing kangaroo mother care (KMC() at the hospital | 12 months
  A pre-defined set of questions will be asked to determine the barriers contributing to practicing kangaroo mother care (KMC) initiation at the hospital. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Number of facilitators to practicing kangaroo mother care (KMC) at the hospital | 12 months
  A pre-defined set of questions will be asked to determine the facilitators contributing to practicing kangaroo mother care (KMC) initiation at the hospital. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Number of barriers to practicing kangaroo mother care (KMC) at home | 12 months
  A pre-defined set of questions will be asked to determine the barriers contributing to practicing kangaroo mother care (KMC) initiation at home. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Number of facilitators to practicing kangaroo mother care (KMC) at home | 12 months
  A pre-defined set of questions will be asked to all the mothers to determine the facilitators contributing to practicing kangaroo mother care (KMC) initiation at home. The Investigators will enroll mothers (n=24), fathers (n=24), and family members (n=24) to undergo in-depth interviews (IDIs).
Percentage of fathers with postpartum depression | 2 weeks, 8 weeks, 6 months, 12 months
  Score on Edinburg Postnatal Depression Scale (EPDS) screening tool obtained by interview with mother. This screening tool is a 10-question tool validated for use among pregnant women in low resource countries. It can be used for screening of perinatal depression, beginning from antenatal period up to 6-8 weeks postnatal age. Each question is scored between 0-3, the highest cumulative score being 30. Cut-off score for fathers with suspected postpartum depression (PPD) will be 9. All fathers who screen 9+ will be categorized to have PPD, all fathers scoring below 9 will be categorized as negative for PPD.
Hours of time father spent with newborn daily | 8 weeks, 6 months, 12 months
  Time (hours/minutes) spent interacting with the newborn/infant each day obtained by interview with the father
Percentage of mothers with depression | 2 weeks, 8 weeks, 6 months, and 12 months
  Patient Health Questionnaire (PHQ-9) is a 9-question patient-administered screening tool for the assessment of depression among mothers and fathers. Since PHQ-9 can be used repeatedly to monitor depressive symptoms among the same patient/study participant, it will be used at different time points throughout the study. The severity scale is as follows:
  1. None: 0-4
  2. Mild: 5-9
  3. Moderate: 10-14
  4. Moderate-Severe: 15-19
  5. Severe: 20-27
Percentage of mothers with self-reported perceived social support | 6 months, 12 months
  Multidimensional Scale of Perceived Social Support (MSPSS) is a tool for screening of perceived social support from family, friends, and significant other.] It, a brief and easy-to-follow self-report measure, is a 12-question tool using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree). It uses positive and negative phrasing to limit response set bias of agreement. Mothers enrolled in the study will be screened using the MSPSS screening tool at 6 and 12 months following enrolment. This total score can also be calculated as a mean score (divide by 12). To calculate the mean subscale scores:
  * Significant Other Subscale: Sum across items 1, 2, 5, & 10, then divide by 4.
  * Family Subscale: Sum across items 3, 4, 8, & 11, then divide by 4.
  * Friends Subscale: Sum across items 6, 7, 9, & 12, then divide by 4.
  Scores are divided into:
  1. Low support: 1 to 2.9
  2. Moderate support: 3 to 5
  3. High support: 5.1 to 7
Cost of admission to kangaroo mother care (KMC) ward | Through KMC discharge of up to 8 weeks
  Government funds spent by the government for admission of one newborn to the kangaroo mother care (KMC) ward per day obtained from government sources. This will estimate the average cost per patient admitted to the KMC ward.
Cost of readmission to the neonatal intensive care unit (NICU) | Through NICU discharge of up to 8 weeks
  Funds spent by the government for readmission of one newborn to the neonatal intensive care unit (NICU) per day obtained from government sources. This will estimate the average cost per patient admitted to the NICU.
Cost associated with hospital readmissions | 12 months
  Funds spent by the government for readmission of one infant to the hospital per day obtained from government sources. This will estimate the average cost per patient readmitted to the hospital.
Out-of-pocket family costs associated with hospital readmissions | 12 months
  Funds spent by the family associated with readmission of one infant to the hospital per day obtained from maternal interview. This will estimate the average funds spent by the family per patient readmitted to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Manasyan, MD, MPH, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Women and Newborn Hospital - University Teaching Hospitals, Lusaka, Lusaka Province, Zambia